CLINICAL TRIAL: NCT00099866
Title: Efficacy and Safety of Vildagliptin Compared to Metformin in Drug Naive Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237A2309
Record Dates: First submitted 2004-12-21; First posted 2004-12-22 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: type 2 diabetes; vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Vildagliptin (Experimental)
  Interventions: Drug: vildagliptin
- Metformin (Active Comparator)
  Interventions: Drug: Metformin Comparator

INTERVENTIONS:
Drug: vildagliptin
  Other Names: LAF237A
  Arms: Vildagliptin
Drug: Metformin Comparator
  Arms: Metformin

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of vildagliptin, an unapproved drug, compared to metformin in lowering overall blood glucose levels in people with type 2 diabetes who have not been previously treated with drug therapy to lower their blood sugar.

ELIGIBILITY:
Inclusion Criteria:

* Not currently on durg therapy for type 2 diabetes
* Body mass index (BMI) in the range 22-45
* Blood glucose criteria must be met

Exclusion Criteria:

* Type 1 diabetes
* Pregnancy or lactation
* Evidence of serious diabetic complications
* Evidence of serious cardiovascular conditions
* Laboratory value abnormalities as defined by the protocol
* Other protocol-defined exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Actual)
Dates: Start 2004-01; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c at 52 weeks

SECONDARY OUTCOMES:
Change from baseline in fasting plasma glucose at 52 weeks
Adverse event profile after 52 weeks of treatment
Change from baseline in body weight at 52 weeks
Change from baseline in fasting lipids at 52 weeks
Change from baseline in HOMA B at 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis investigative Site, Investigative Sites, Germany

REFERENCES:
- [Derived] Gnesin F, Thuesen ACB, Kahler LKA, Madsbad S, Hemmingsen B. Metformin monotherapy for adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Jun 5;6(6):CD012906. doi: 10.1002/14651858.CD012906.pub2. PMID 32501595
- [Derived] Pratley RE, Schweizer A, Rosenstock J, Foley JE, Banerji MA, Pi-Sunyer FX, Mills D, Dejager S. Robust improvements in fasting and prandial measures of beta-cell function with vildagliptin in drug-naive patients: analysis of pooled vildagliptin monotherapy database. Diabetes Obes Metab. 2008 Sep;10(10):931-8. doi: 10.1111/j.1463-1326.2007.00835.x. Epub 2007 Dec 17. PMID 18093207
- [Derived] Pratley RE, Rosenstock J, Pi-Sunyer FX, Banerji MA, Schweizer A, Couturier A, Dejager S. Management of type 2 diabetes in treatment-naive elderly patients: benefits and risks of vildagliptin monotherapy. Diabetes Care. 2007 Dec;30(12):3017-22. doi: 10.2337/dc07-1188. Epub 2007 Sep 18. PMID 17878242